CLINICAL TRIAL: NCT00353080
Title: A Two-year, Multicenter, Double-blind, Randomized, Placebo-controlled and Parallel Group Study of Oral Risedronate 5 mg Daily in the Prevention of Osteoporosis in Osteopenic Postmenopausal Women (More Than 5 Years Postmenopausal)
Brief Title: Risedronate In The Prevention Of Osteoporosis In Osteopenic Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Procter and Gamble (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EFC6064; HMR4003B/3001
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Prevention of postmenopausal osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: risedronate (HMR4003)

SUMMARY:
To confirm the superiority of 5 mg daily risedronate as compared to placebo in maintaining or increasing bone mass in lumbar spine in osteopenic postmenopausal women

To confirm the efficacy of 5 mg daily risedronate in osteopenic postmenopausal women in maintaining or increasing bone mass in proximal femur and decreasing bone resorption

To confirm general safety of 5 mg daily risedronate as compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, healthy postmenopausal women with

  * Natural menopause and more than 5 years after their last menstrual period
  * or surgical menopause and more than 5 years after surgery
  * osteopenia (lumbar spine T score between 1 and 2.5 SD below the mean value in normal young women).
* With at least one risk factor for osteoporosis

Exclusion Criteria:

* Women who have received hormone replacement therapy (with estrogen and/or progestogen and/or androgen) or raloxifene within 3 months before visit 2 or calcitonin or calcitriol within 4 weeks before visit 2

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2002-12; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Percent changes from baseline in lumbar spine bone mineral density (BMD) at Month 24 measured by DXA.

SECONDARY OUTCOMES:
Percent changes in proximal femur BMD from baseline at month 12 and 24 (DXA)
Percent of responders (subjects with a positive change in lumbar spine BMD from baseline)at Month 12 and 24
Percent changes in bone turnover markers after 12 and 24 months of treatment
Physical examination and hematology tests before and after 12 and 24 months of treatment;Serum Chemistry before and after 6, 12 and 24 months of treatment
Occurrence of adverse events at each visit with special interest for upper gastro-intestinal events

CONTACTS AND LOCATIONS:
Overall Officials: Välimäki Matti, MD, Principal Investigator — Division of Endocrinology, Helsinki University Central Hospital, Helsinki, Finland
Locations (5):
- Sanofi-Aventis, Helsinki, Finland
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Oslo, Norway
- Sanofi-Aventis, Madrid, Spain
- Sanofi-Aventis, Stockholm, Sweden

REFERENCES:
- [Result] Valimaki MJ, Farrerons-Minguella J, Halse J, Kroger H, Maroni M, Mulder H, Munoz-Torres M, Saaf M, Snorre Ofjord E. Effects of risedronate 5 mg/d on bone mineral density and bone turnover markers in late-postmenopausal women with osteopenia: a multinational, 24-month, randomized, double-blind, placebo-controlled, parallel-group, phase III trial. Clin Ther. 2007 Sep;29(9):1937-49. doi: 10.1016/j.clinthera.2007.09.017. PMID 18035193